CLINICAL TRIAL: NCT04140305
Title: A Multicenter, Longitudinal, Open-Label, Single-Arm Study Describing Cognitive Processing Speed Changes in Relapsing Multiple Sclerosis Subjects Treated With Ozanimod (RPC-1063)
Brief Title: Study Describing Cognitive Processing Speed Changes in Relapsing Multiple Sclerosis Subjects Treated With Ozanimod (RPC-1063)
Acronym: ENLIGHTEN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business objective has changed
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RPC-1063-MS-001; U1111-1240-5667 (Other: WHO)
Record Dates: First submitted 2019-10-24; First posted 2019-10-25 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; RPC-1063; Ozanimod; Phase 3b
MeSH Terms: conditions — Multiple Sclerosis | interventions — ozanimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administration of RPC-1063 (Experimental): Patients with relapsing MS will receive RPC-1063 orally:
  Interventions: Drug: RPC-1063

INTERVENTIONS:
Drug: RPC-1063 — Oral capsule
  Other Names: Ozanimod

SUMMARY:
This is a multicenter, longitudinal, single-arm, open-label study to describe the change from baseline in cognitive processing speed, measured by the SDMT, in subjects with RMS treated with ozanimod HCl 1 mg at 3 years.

All subjects will receive orally administered ozanimod HCl 1 mg. The primary efficacy endpoint is the proportion of subjects with a clinically meaningful increase in raw score of ≥ 4 points or 10% from baseline (improved). The treatment period is 36 months. For all subjects who finish the subject and for those who discontinue, there will be a 30-day (± 15 days) and a 90-day (± 10 days) Safety Follow-up Visit. There is no planned protocol extension following the end of the study. Approximately 250 subjects with RMS will be recruited for this study.

Subjects with RMS will be enrolled in this study if they have received ≤ 1 DMT, have an EDSS ≤ 3.5, and have been diagnosed with RMS within 5 years of study entry. The Investigator will be responsible for the overall conduct of the study at the site, confirmation of subject eligibility, routine study subject clinical management including for MS relapses, and management of AEs.

ELIGIBILITY:
Inclusion Criteria:

Below are some criteria for inclusion. Additional Inclusion criteria apply.

1. Subject must understand and voluntarily sign an informed consent form (ICF) prior to any study-related assessments/procedures being conducted.
2. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
3. Subject is male or female 18 to 65 years of age (inclusive) at the time of signing of the ICF.
4. Subject has a diagnosis of MS according to the 2010 or 2017 Revised McDonald criteria.
5. Subjects has ≤ 5 years since time of RMS diagnosis.
6. Subject has ≤ 1 approved RMS DMT at time of study entry.

Exclusion Criteria:

Following are some criteria that would exclude the subject from participation. Additional exclusion criteria apply.

Exclusions Related to General Health

1. Subject has any clinically relevant hepatic, neurological, pulmonary, ophthalmological, endocrine, psychiatric, or other major systemic disease making implementation of the protocol or interpretation of the study difficult or that would put the subject at risk by participating in the study. Subjects with mild or moderate asthma, and subjects with other mild pulmonary disease (eg, chronic obstructive pulmonary disease [COPD]) may be included in the study.
2. Subject has a presence of other neurologic disorders to explain the progressive neurologic disability (as defined in the key inclusion criteria) or that might affect cognition.
3. Subject has a visual or other sensorimotor impairment likely to confound test performance.
4. Subject has a presence of > 10 GdE lesions on the Baseline brain MRI scan.
5. Subject has a history of developmental disorder (eg, attention-deficit/hyperactivity disorder [ADHD], learning disability).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with an increase in raw score of ≥ 4 points or 10% from baseline (improved) | Up to approximately 3 years
  Symbol Digit Modalities Test

SECONDARY OUTCOMES:
Proportion of subjects with a decrease in raw score of ≥ 4 points or 10% from baseline (worsened) | Up to approximately 3 years
  Symbol Digit Modalities Test
Proportion of subjects with a raw score change from baseline who do not meet the improved or worsened definition (stable) | Up to approximately 3 years
  Symbol Digit Modalities Test
Proportion of subjects with an increase in raw score of ≥ 3 points from baseline | Up to approximately 3 years
  Symbol Digit Modalities Test
Proportion of subjects with a decrease in raw score of ≥ 3 points from baseline | Up to approximately 3 years
  Symbol Digit Modalities Test
Change from baseline in Symbol Digit Modalities Test (SMDT) | Up to approximately 3 years
  The SDMT is a measure of cognitive processing speed
Percent change from baseline in thalamic, cortical grey matter, whole brain, lateral ventricular, and MOV volumes | Up to approximately 3 years
  Magnetic resonance imaging (MRI) brain volume
Proportion of subjects free of gadolinium enhancing (GdE) lesions over 3 years | Up to approximately 3 years
  Magnetic Resonance Imaging
GdE lesion volume over 3 years | Up to approximately 3 years
  Magnetic Resonance Imaging
Number of unique new or enlarging hyperintense T2-weighted lesions and their volume from baseline to Year 3 | Up to approximately 3 years
  Magnetic Resonance Imaging
Number of unique new or enlarging hypointense T1 weighted lesions and their volume from baseline to Year 3 | Up to approximately 3 years
  Magnetic Resonance Imaging
Treatment Satisfaction Questionnaire for Medication (TSQM v1.4) | Up to approximately 3 years
  Change is TSQM score over 3 years
Work Productivity and Activity Impairment-Multiple Sclerosis (WPAI-MS) | Up to approximately 3 years
  Change in WPAI score over 3 years
Fatigue Severity Scale (FSS) | Up to approximately 3 years
  The Fatigue Severity Scale (FSS) questionnaire contains nine statements that attempt to explore severity of fatigue symptoms.
Multiple Sclerosis Quality of Life-54 (MSQOL-54) | Up to approximately 3 years
  The MSQOL-54 is a multidimensional health-related QOL measure that combines both generic and MS-specific items into a single instrument
Hospital Anxiety and Depression Scale (HADS) | Up to approximately 3 years
  The HADS was developed to identify anxiety disorders and depression among subjects in nonpsychiatric hospital clinics
Annualized relapse rate (ARR) | Up to approximately 3 years
  Change in relapse rate over 3 years
Timed 25-foot Walk (T25W) | Up to approximately 3 years
  Disability progression assessed by 20% worsening from baseline over 3 years on T25W
Nine-hole Peg Test (9-HPT) | Up to approximately 3 years
  Change from baseline in the time in seconds needed to complete test activity
Expanded Disability Status Scale (EDSS) | Up to approximately 3 years
  Change from baseline in EDSS score (0-10) yearly and at 3 years
Adverse Events (AEs) | Up to approximately 3 years
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a pre-existing condition) should be considered an AE.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (61):
- United States (56):
  - Local Institution - 123, Birmingham, Alabama
  - Local Institution - 136, Cullman, Alabama
  - Local Institution - 153, Mobile, Alabama
  - Local Institution - 162, Phoenix, Arizona
  - Local Institution - 128, Pasadena, California
  - Local Institution - 164, Sacramento, California
  - Local Institution - 107, Aurora, Colorado
  - Local Institution - 102, Colorado Springs, Colorado
  - Local Institution - 144, Fort Collins, Colorado
  - Local Institution - 109, Washington D.C., District of Columbia
  - Local Institution - 140, Boca Raton, Florida
  - Local Institution - 158, Vero Beach, Florida
  - Local Institution - 114, Savannah, Georgia
  - Northwest Neurology, Ltd, Hoffman Estates, Illinois
  - Local Institution - 108, Northbrook, Illinois
  - Local Institution - 148, Fort Wayne, Indiana
  - Local Institution - 126, Ames, Iowa
  - Local Institution - 173, Kansas City, Kansas
  - Local Institution - 133, Alexandria, Louisiana
  - Local Institution - 152, Detroit, Michigan
  - Local Institution - 112, Detroit, Michigan
  - Local Institution - 122, St Louis, Missouri
  - Local Institution - 143, St Louis, Missouri
  - Advanced Neurology Specialists, Great Falls, Montana
  - Local Institution - 149, Teaneck, New Jersey
  - Dent Neurologic Institute, Amherst, New York
  - Local Institution - 137, Buffalo, New York
  - Local Institution - 160, East Setauket, New York
  - Local Institution - 130, New York, New York
  - Local Institution - 121, New York, New York
  - Local Institution - 146, Patchogue, New York
  - Local Institution - 131, Chapel Hill, North Carolina
  - Local Institution - 106, Greensboro, North Carolina
  - Local Institution - 170, Mooresville, North Carolina
  - Raleigh Neurology Associates PA, Raleigh, North Carolina
  - Local Institution - 174, Cincinnati, Ohio
  - Local Institution - 171, Cleveland, Ohio
  - Local Institution - 142, Dayton, Ohio
  - Local Institution - 157, Oklahoma City, Oklahoma
  - Local Institution - 159, Philadelphia, Pennsylvania
  - Local Institution - 169, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Local Institution - 125, Franklin, Tennessee
  - Local Institution - 119, Knoxville, Tennessee
  - Local Institution - 139, Dallas, Texas
  - Local Institution - 113, Round Rock, Texas
  - Local Institution - 101, San Antonio, Texas
  - Local Institution - 103, Norfolk, Virginia
  - Local Institution - 141, Kirkland, Washington
  - Local Institution - 168, Seattle, Washington
  - Local Institution - 172, Spokane, Washington
  - Local Institution - 124, Tacoma, Washington
  - Local Institution - 156, Huntington, West Virginia
  - Local Institution - 150, Morgantown, West Virginia
  - Local Institution - 167, Madison, Wisconsin
  - Local Institution - 147, Milwaukee, Wisconsin
- Canada (4):
  - Local Institution - 203, London, Ontario
  - Local Institution - 204, Ottawa, Ontario
  - Local Institution - 206, Montreal, Quebec
  - Local Institution - 207, Halifax
- Local Institution - 166, Guaynabo, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com